CLINICAL TRIAL: NCT04639661
Title: Predictors of Periodontal Outcomes in Patients 5 to 10 Years Post-sanative Therapy
Brief Title: Predictors of Periodontal Outcomes Post-sanative Therapy
Status: Terminated | Type: Observational
Why Stopped: Challenges with recruiting patients during the COVID-19 pandemic.
Sponsor: Brock University (Other)
Collaborators: Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor, Brock University
Other Study IDs: 20-070
Record Dates: First submitted 2020-11-09; First posted 2020-11-20 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Periodontal Diseases; Periodontal Pocket
Keywords: Periodontal therapy; Flavonoids; Tea; Dietary intake; Supplements; Physical activity; Exercise; Sedentary time; Estrogen; Lifetime estrogen exposure; Periodontal maintenance
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Periodontal disease is a chronic inflammatory disease of the tissues surrounding the teeth and is one of the leading causes of tooth loss. Sanative therapy (ST) is a non-surgical procedure that allows for removal of bacteria from the deep pockets that form around teeth and is the frontline treatment for periodontal disease. Post-ST, patients require ongoing maintenance appointments to maintain their oral health, though whether risk factors for periodontal disease remain a predictor of periodontal health post-ST has not been comprehensively investigated. Risk factors to be examined include physical activity, exercise, sedentary time, flavonoid intake, protein intake, BMI, sex, age, smoking status, and number of sites with periodontal probing depth (PPD) ≥ 4mm at baseline.

DETAILED DESCRIPTION:
Periodontal disease is a main cause of tooth loss. Patients with periodontal disease may receive sanative therapy (ST), a deep cleaning of the teeth that helps prevent the progression of periodontal disease. Post-ST, maintenance appointments are an important part of the strategy used to help these patients prevent the progression of periodontal disease and maintain their periodontal health. Given that numerous chronic diseases, obesity, low levels of physical activity, being a smoker, poor diet, and older age are all risk factors for periodontal disease, these factors may also be predictive of worse periodontal health 5 to 10 years post-ST. Many modifiable periodontal risk factors such a physical activity, exercise, and obesity have not been studied in relation to periodontal outcomes post-ST, and other factors such as diet, sex and age have not been comprehensively studied. The primary objective of this study is to determine, at 5 to 10 years post-ST, if physical activity, exercise, sedentary time, flavonoid intake, protein intake, BMI, sex, age, smoking status, and number of sites with periodontal probing depth (PPD) ≥ 4 mm at baseline are significant predictors of periodontal health. A secondary objective is to determine if lifetime estrogen exposure impacts periodontal health in women. Periodontal health will be measured using probing depth, tooth loss, bleeding on probing and plaque index. Established questionnaires will be used to assess dietary intake, physical activity and sedentary behaviour. Within the study the investigators will also assess if and how a patient's periodontal health has been impacted by clinic closures and rescheduling of maintenance appointments that were mandated by regulatory organizations as a result of the COVID-19 pandemic. The investigators will also ask questions about changes in diet, physical activity and oral hygiene during COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone sanative therapy (ST) in the past 5 to 10 years
* Age > 19 years
* Willingness and ability to provide informed consent. Participants must be able and willing to complete online questionnaires from home and give permission for access to their periodontal records from the time of their sanative therapy to present day

Exclusion Criteria:

* Individuals with physical or mental limitations that inhibit them from conducting their own personal oral hygiene (oral hygiene is a key component in maintaining periodontal health)
* Women who are currently pregnant or breastfeeding (hormonal changes during pregnancy are known to cause gingival inflammation)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent sanative therapy to manage periodontal disease at this clinic 5 to 10 years before present-day appointment. Only patients who have maintained regular maintenance appointments after receiving sanative therapy will be eligible.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Probing depth | At maintenance appointment (present day)
  This is a routine clinical measure of periodontal health (measured in mm)
Probing depth | Pre-sanative therapy
  This is a routine clinical measure of periodontal health (measured in mm)
Probing depth | 8-12 weeks post-sanative therapy
  This is a routine clinical measure of periodontal health (measured in mm)
Bleeding on probing | At maintenance appointment (present day) and retrospectively from the clinical record from the time of sanative therapy (5 to 10 years ago) onwards
  This is a clinical measure of inflammation and represented as the percent of bleeding sites that are measured at 6 sites per tooth
Bleeding on probing | Pre-sanative therapy
  This is a clinical measure of inflammation and represented as the percent of bleeding sites that are measured at 6 sites per tooth
Bleeding on probing | 8-12 weeks post-sanative therapy
  This is a clinical measure of inflammation and represented as the percent of bleeding sites that are measured at 6 sites per tooth

SECONDARY OUTCOMES:
Tooth Loss | At maintenance appointment (present day) and retrospectively from the clinical record from the time of sanative therapy (5 to 10 years ago) onwards
  Will be measured as the number of teeth lost due to periodontal disease
Tooth Loss | Pre-sanative therapy
  Will be measured as the number of teeth lost due to periodontal disease
Tooth Loss | 8-12 weeks post-sanative therapy
  Will be measured as the number of teeth lost due to periodontal disease
O'Leary Index of Plaque Control | At maintenance appointment (present day) and retrospectively from the clinical record from the time of sanative therapy (5 to 10 years ago) onwards
  The patient's plaque index= the number of plaque-containing surfaces divided by the total number of available surfaces. The minimum plaque index would be 0% which represents no tooth surfaces that contain plaque/ The maximum plaque index would be 100%, which represents all surfaces of the patient's teeth containing plaque.
O'Leary Index of Plaque Control | Pre-sanative therapy
  The patient's plaque index= the number of plaque-containing surfaces divided by the total number of available surfaces. The minimum plaque index would be 0% which represents no tooth surfaces that contain plaque/ The maximum plaque index would be 100%, which represents all surfaces of the patient's teeth containing plaque.
O'Leary Index of Plaque Control | 8-12 weeks post-sanative therapy
  The patient's plaque index= the number of plaque-containing surfaces divided by the total number of available surfaces. The minimum plaque index would be 0% which represents no tooth surfaces that contain plaque/ The maximum plaque index would be 100%, which represents all surfaces of the patient's teeth containing plaque.

OTHER OUTCOMES:
Body Mass Index (BMI) | Patients will complete this in an online questionnaire at present day (baseline).
  Patients will self-report their height and weight in an online questionnaire. This information will be used to calculate BMI which is a known risk factor of periodontal disease.
Godin Leisure Time Exercise Questionnaire | Patients will complete this in an online questionnaire at present day (baseline).
  This questionnaire measures, at one time point, self-reported exercise habits for the past 7 days. This questionnaire includes 4 items and has been combined with the International Physical Activity Questionnaire.
  Name of score: Weekly leisure activity score; Minimum score: 0 units and Maximum score: 24 units or more and defined as "active". A higher score indicates a better outcome.
International Physical Activity Questionnaire (IPAQ) | Patients will complete this online questionnaire at present day (baseline).
  This questionnaire measures, at one time point, self-reported physical activity and sedentary behavior habits. It contains 27 items and has been combined with the Godin Leisure Time Exercise Questionnaire and modified version of the indices of estrogen exposure questionnaire in an online format. They will self-report their physical activity and sedentary behavior for the past 7 days.
  Name of score: Weekly physical activity score; Minimum score: 1 and defined as "low physical activity" and Maximumscore: 3 and defined as "high physical activity". A higher score indicates a better outcome.
Flavonoid and protein intake | Patients will report their dietary intake at present day (baseline) for the past 24 hours. This will be done three times for three separate dates.
  Flavonoid and protein intake will be measured with the automated self-administered dietary intake (ASA-24) questionnaire. This is an online food recall that patients will complete three times, reporting on their dietary intake from the last 24 hours.
Lifetime estrogen exposure (LEE) | Patients will complete this online questionnaire at present day (baseline).
  The indices of estrogen exposure questionnaire will be used to determine LEE using the estimated lifetime estrogen exposure (ELEE) model. The ELEE reflects the reproductive span, comprising a woman's time between age at menarche and age at menopause (or age at recruitment minus age at menarche for pre-menopausal women) minus 1 year for each pregnancy and duration of breastfeeding, calculated at the time at recruitment.
Dietary supplement and tea intake | Patients will complete this questionnaire online prior to their maintenance appointment
  Intakes of specific dietary supplements and tea will be measured using a dietary supplement and tea intake questionnaire.
COVID-19 Interview questions | Patients will complete these interview questions during their one-on-one virtual meeting with a member of the research team at present day (baseline).
  Patients will be asked interview questions about changes to their dietary intake, physical activity and oral hygiene habits resulting from the COVID-19 pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Wendy E Ward, PhD, Principal Investigator — Brock University
Locations (2):
- Canada (2):
  - Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery, Fonthill, Ontario
  - Brock University, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: Undecided